CLINICAL TRIAL: NCT06501859
Title: Rehabilitation With the Shoulder Pacemaker After Reverse Shoulder Arthroplasty
Brief Title: Rehabilitation With the Shoulder Pacemaker
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Joyce, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 163105
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Injuries
Keywords: Reverse Shoulder Arthroplasty (RSA); Shoulder Pacemaker; Rehabilitation; Range of motion; Pain
MeSH Terms: conditions — Shoulder Injuries; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of care physical therapy (Active Comparator): Control group and will not use the shoulder pacemaker, but will participate in a standardized physical therapy protocol for 3 months.
  Interventions: Other: Standard of care physical therapy
- Shoulder pacemaker with physical therapy (Experimental): Include a standardized physical therapy protocol with utilization of the Shoulder Pacemaker device 3 times per week over a 3-month period starting at 6 weeks post-operatively.
  Interventions: Device: Shoulder pacemaker with physical therapy

INTERVENTIONS:
Other: Standard of care physical therapy — Standard rehabilitation protocol for 3 months.
  Arms: Standard of care physical therapy
Device: Shoulder pacemaker with physical therapy — Standardized rehabilitation protocol with utilization of the shoulder pacemaker device 3 times per week over a 3-month period.
  Arms: Shoulder pacemaker with physical therapy

SUMMARY:
The investigators purpose of the proposed study is to use the FDA approved Shoulder Pacemaker device in patients undergoing reverse shoulder arthroplasty and study the functional outcomes compared to a standard post-operative rehabilitation program. The investigators hypothesize that use of the Shoulder Pacemaker reduce pain and will allow for improved range of motion and function in patients undergoing RSA. The findings of this research may very well improve function in RSA patients through a novel, non-invasive approach.

DETAILED DESCRIPTION:
The reverse shoulder arthroplasty (RSA) has increased utility in recent years for shoulder conditions such as rotator cuff tear arthropathy, massive irreparable rotator cuff tears, severe glenohumeral arthritis, proximal humerus fracture, and failed shoulder arthroplasty. While RSA may commonly be the only surgical treatment for some of these conditions, the outcomes and adverse event profiles are significant. Specifically, RSA patients often complain of poor range of motion and function with the arm above the head. Despite many attempts at solving these shortcomings with new implant design iterations and improved implant positioning, these continue to be a source of frustration with patients and surgeons alike.

Poor scapulothoracic motion is associated with poor shoulder range of motion, especially after RSA. Past investigators have shown that in certain RSA patients, there is a near complete loss of glenohumeral motion and forward elevation and abduction is highly dependent on scapulothoracic motion. In a separate study, In addition, these investigators demonstrated that internal rotation after RSA is largely dependent on scapulothoracic motion. Several years ago, a device called the Shoulder Pacemaker (Alyve Medical, Denver, CO) was developed initially for the treatment of functional instability in the setting of scapular dyskinesis. It functions as a wearable muscle electrostimulator that allows for periscapular muscle stimulation as well as feedback on shoulder range of motion. The motion technology recognizes muscle movement and automatically sets the appropriate stimulation intensity according to the movement. This improves scapular muscle recruitment during range of motion. While the data is limited, there has been some early promising results for this pathology. As function after RSA is particularly reliant on scapulothoracic function, the current investigators may infer that use of the Shoulder Pacemaker device may function well in patients with reverse shoulder replacements. Specifically, the device would allow patients to train their periscapular musculature after RSA to improve global shoulder motion and function. To the current investigators knowledge, there is no current research on the use of the Shoulder Pacemaker after RSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for primary reverse shoulder arthroplasty
* Surgery at University of Utah Facilities
* Patients between the ages 18-80.

Exclusion Criteria:

* Prior ipsilateral shoulder arthroplasty
* Inability or unwillingness to participate in the rehabilitation protocol
* Prior cardiac pacemaker or spinal cord stimulator
* Age over 80
* History of periscapular surgery
* History of ipsilateral neurologic injury
* Prisoners
* Patients requiring prolonged immobilization deviating from standard protocol
* Patients who have an implantable medical device or other electrical device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons score | Pre-operatively
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 6 weeks after surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 3 months after surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 6 months after surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.
American Shoulder and Elbow Surgeons score | 1 year after surgery
  Shoulder specific scoring system out of 100. A patient-reported score with visual analog scale for pain and functional subscales ranging from 0 (worse pain and function loss) to 50 (no pain and excellent function). Both scores are summed for a maximum score of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Joyce, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States